CLINICAL TRIAL: NCT01277718
Title: A Phase 1, Open-Label, 3-Period, Randomized, Crossover Study to Evaluate the Effect of a Proton-Pump Inhibitor (Rabeprazole) on the Relative Bioavailability of GDC-0973 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of a Proton-Pump Inhibitor (Rabeprazole) on the Relative Bioavailability of Cobimetinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MEK4954g
Record Dates: First submitted 2011-01-07; First posted 2011-01-17 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — cobimetinib; Rabeprazole

ARMS (2):
- Treatment A first, then Treatment B, followed by Treatment C (Experimental): Treatment A in Period 1: One 20-mg tablet of cobimetinib will be administered orally with 240 milliliters (mL) room temperature water after at least an 8-hour fast. Treatment B in Period 2: 20 mg oral rabeprazole will be administered once daily for 4 days starting on Day -4. On Day 1, 20 mg rabeprazole will be administered in fasted state followed by one 20-mg tablet of cobimetinib administration orally with 240 mL room temperature water after at least an 8-hour fast. Treatment C in Period 3: 20 mg oral rabeprazole will be administered once daily for 4 days starting on Day -4. On Day 1, 20 mg rabeprazole will be administered in fasted state. Approximately 30 minutes later, participants will be provided a standardized Food and Drug Administration (FDA) high-fat meal, and approximately 30 minutes after starting meal, one 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water. There will be a 13-day washout between cobimetinib doses of each period.
  Interventions: Drug: Cobimetinib; Drug: Rabeprazole
- Treatment A first, then Treatment C, followed by Treatment B (Experimental): Treatment A in Period 1: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast. Treatment C in Period 2: 20 mg oral rabeprazole will be administered once daily for 4 days starting on Day -4. On Day 1 of the treatment period, 20 mg rabeprazole will be administered in fasted state. Approximately 30 minutes later, participants will be provided a standardized FDA high-fat meal, and approximately 30 minutes after starting meal, one 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water. Treatment B in Period 3: 20 mg oral rabeprazole will be administered once daily for 4 days starting on Day -4. On Day 1 of treatment period, 20 mg rabeprazole will be administered in fasted state followed by one 20-mg tablet of cobimetinib administration orally with 240 mL room temperature water after at least an 8-hour fast. There will be a 13-day washout between cobimetinib doses of each period.
  Interventions: Drug: Cobimetinib; Drug: Rabeprazole

INTERVENTIONS:
Drug: Cobimetinib — One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast or approximately 30 minutes after starting the standardized FDA high-fat meal.
  Other Names: GDC-0973; XL518
Drug: Rabeprazole — Rabeprazole 20 mg will be administered orally once daily for 4 days starting on Day -4 and on Day 1 of the treatment period.

SUMMARY:
This is a Phase 1, single-center, open-label, randomized, 3-period, 2-sequence crossover study of cobimetinib in healthy participants to evaluate the effect of the proton-pump inhibitor (PPI) rabeprazole on the relative bioavailability of cobimetinib in healthy participants when administered in the fed or fasted states.

ELIGIBILITY:
Inclusion Criteria

* With a body mass index range of 18.5 to 29.9 kilograms per meter square (kg/m^2)
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), and vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory
* Negative test for selected drugs of abuse at Screening (does not include alcohol) and at each Check-in
* Negative hepatitis panel (including hepatitis B virus surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]) and negative human immunodeficiency virus (HIV) antibody screens
* Healthy males and females of nonchildbearing potential who agree to use effective contraception

Exclusion Criteria

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs, except that appendectomy, hernia repair, and/or cholecystectomy will be allowed
* History or presence of an abnormal ECG
* History of alcoholism or drug addiction within 1 year prior to Period 1 Check-in
* Use of any tobacco- or nicotine-containing products within 6 months prior to Period 1 Check-in
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days or 5 half-lives, whichever is longer, prior to Period 1 Check-in
* Use of any prescription medications/products within 14 days prior to Period 1 Check-in
* Use of any over-the-counter, non-prescription preparations within 7 days prior to Period 1 Check-in
* Use of alcohol-, grapefruit-, or caffeine-containing foods or beverages within 72 hours prior to Period 1 Check-in
* Poor peripheral venous access
* Any acute or chronic condition that would limit the participant's ability to complete and/or participate in this clinical study
* Female participant is pregnant, lactating, or breastfeeding
* Use of PPIs or histamine H2 receptor antagonists within 1 month prior to Period 1 Check-in
* Known hypersensitivity to rabeprazole or any of its components or to derived products of benzimidazoles
* Predisposing factors to retinal vein occlusion (RVO)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Rooney, M.D., PhD, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A First, Then Treatment B, Followed by Treatment C: Treatment A in Period 1: One 20-mg tablet of cobimetinib administered orally with 240 milliliters (mL) room temperature water after at least an 8-hour fast. Treatment B in Period 2: 20 mg oral rabeprazole administered once daily for 4 days starting on Day -4. On Day 1 of the treatment period, 20 mg rabeprazole was administered in fasted state followed by one 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast. Treatment C in Period 3: 20 mg oral rabeprazole administered once daily for 4 days starting on Day -4. On Day 1, 20 mg rabeprazole was administered in fasted state. Approximately 30 minutes later, participants were provided a standardized Food and Drug Administration (FDA) high-fat meal, and approximately 30 minutes after starting the meal, one 20-mg tablet of cobimetinib was administered orally with 240 mL room temperature water. There was minimum of a 13-day washout between cobimetinib doses of each period.
- Treatment A First, Then Treatment C, Followed by Treatment B: Treatment A in Period 1: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast. Treatment C in Period 2: 20 mg oral rabeprazole administered once daily for 4 days starting on Day -4. On Day 1 of the treatment period, 20 mg rabeprazole was administered in fasted state. Approximately 30 minutes later, participants were provided a standardized FDA high-fat meal, and approximately 30 minutes after starting the meal, one 20-mg tablet of cobimetinib was administered orally with 240 mL room temperature water. Treatment B in Period 3: 20 mg oral rabeprazole administered once daily for 4 days starting on Day -4. On Day 1 of the treatment period, 20 mg rabeprazole was administered in fasted state followed by one 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast. There was minimum of a 13-day washout between cobimetinib doses of each period.
Period: Period 1 - First Intervention
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period of 13 Days
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2 - Second Intervention
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B
Started | 10 | 10
Completed | 10 | 7
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 2
Period: Washout Period of 13 Days
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0
Period: Period 3 - Third Intervention
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Entire Study Population: All participants randomized to any treatment.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 31 [22 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Cobimetinib
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Time Frame: Day 1 at 0 hour (predose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 hours postdose
Population: Pharmacokinetic parameters populations included all enrolled participants. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Groups:
- Cobimetinib [Fasted]: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast.
- Cobimetinib [Fasted] + Rabeprazole: Participants received 20 mg oral rabeprazole once daily for 4 days starting on Day -4. On Day 1 of the treatment period, 20 mg rabeprazole was administered in fasted state followed by one 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast.
- Cobimetinib [Fed] + Rabeprazole: Participants received 20 mg oral rabeprazole once daily for 4 days starting on Day -4. On Day 1 of the treatment period, 20 mg rabeprazole was administered in fasted state. Approximately 30 minutes later, participants were provided a standardized FDA high-fat meal, and approximately 30 minutes after starting the meal, one 20-mg tablet of cobimetinib was administered orally with 240 mL room temperature water.
Arm/Group | Cobimetinib [Fasted] | Cobimetinib [Fasted] + Rabeprazole | Cobimetinib [Fed] + Rabeprazole
Number analyzed (Participants) | 20 | 16 | 17
nanograms*hours/milliliter (ng*hr/mL) | 778 (32.8) | 864 (39.1) | 846 (48.2)
Statistical Analysis 1: Comparison: Cobimetinib [Fasted] vs Cobimetinib [Fasted] + Rabeprazole; Test type: Superiority or Other; Ratio of Least Squares (LS) Means (in %) = 111, 90% CI 2-sided [98.02 to 124.99] — LS mean was calculated from Analysis of variance (ANOVA). Data for AUCinf were natural log-transformed prior to analysis. Ratio of AUCinf LS means for log-transformed parameter (expressed as a percent)
Statistical Analysis 2: Comparison: Cobimetinib [Fasted] + Rabeprazole vs Cobimetinib [Fed] + Rabeprazole; Test type: Superiority or Other; Ratio of LS Means (in %) = 96.2, 90% CI 2-sided [85.06 to 108.77] — LS mean was calculated from ANOVA. Data for AUCinf were natural log-transformed prior to analysis. Ratio of AUCinf LS means for log-transformed parameter (expressed as a percent)
Statistical Analysis 3: Comparison: Cobimetinib [Fasted] vs Cobimetinib [Fed] + Rabeprazole; Test type: Superiority or Other; Ratio of LS Means (in %) = 106, 90% CI 2-sided [94.53 to 119.91] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Maximum Observed Concentration of Cobimetinib
Time Frame: Day 1 at 0 hour (predose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cobimetinib [Fasted] | Cobimetinib [Fasted] + Rabeprazole | Cobimetinib [Fed] + Rabeprazole
Number analyzed (Participants) | 20 | 17 | 17
nanograms per milliliter (ng/mL) | 17.0 (35.3) | 17.2 (36.0) | 14.8 (51.2)
Statistical Analysis 1: Comparison: Cobimetinib [Fasted] vs Cobimetinib [Fasted] + Rabeprazole; Test type: Superiority or Other; Ratio of LS Means (in %) = 100, 90% CI 2-sided [85.09 to 118.03] — LS mean was calculated from ANOVA. Data for Cmax were natural log-transformed prior to analysis. Ratio of Cmax LS means for log-transformed parameter (expressed as a percent)
Statistical Analysis 2: Comparison: Cobimetinib [Fasted] + Rabeprazole vs Cobimetinib [Fed] + Rabeprazole; Test type: Superiority or Other; Ratio of LS Means (in %) = 85.7, 90% CI 2-sided [72.51 to 101.33] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Cobimetinib [Fasted] vs Cobimetinib [Fed] + Rabeprazole; Test type: Superiority or Other; Ratio of LS Means (in %) = 85.9, 90% CI 2-sided [72.94 to 101.17] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from start of study treatment in first period to end of last period (up to 36 days)
Description: Three participants discontinued study in second period and did not receive Cobimetinib [Fasted] + Rabeprazole in third period. Therefore, only 17 participants were evaluable for adverse events in the Cobimetinib [Fasted] + Rabeprazole treatment arm.
Arm/Group | Cobimetinib [Fasted] | Cobimetinib [Fasted] + Rabeprazole | Cobimetinib [Fed] + Rabeprazole
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 10/17 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cobimetinib [Fasted] (N=20) | Cobimetinib [Fasted] + Rabeprazole (N=17) | Cobimetinib [Fed] + Rabeprazole (N=20)
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract Infection (Infections and infestations) | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 1 | 0
Scleral hyperaemia (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.